CLINICAL TRIAL: NCT05355259
Title: ACCESS : ACtive Catheterization for EndovaScular TreatmentS
Brief Title: ACtive Catheterization for EndovaScular TreatmentS
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basecamp Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCV-FIH-001
Record Dates: First submitted 2022-04-20; First posted 2022-05-02 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Unruptured Intracranial Aneurysm; Arteriovenous Cerebral Malformations; Carotid Stenosis
Keywords: Active catheterization / guidewire; Endovascular treatments
MeSH Terms: conditions — Intracranial Arteriovenous Malformations; Carotid Stenosis

STUDY DESIGN:
Intervention Model Description: This is a prospective monocenter, non-randomized, open clinical investigation to evaluate the safety and technical success of the Basecamp Vascular controllable directional GECKO guidewire when used to facilitate endovascular access to the targeted vessel in order to treat the vascular lesion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GECKO Active Guidewire Use (Experimental): All patients will be treated using the GECKO guidewire to facilitate endovascular access to the targeted vessel in order to treat the vascular lesion.
  Interventions: Device: GECKO Active Guidewire

INTERVENTIONS:
Device: GECKO Active Guidewire — The GECKO device is intended to introduce devices used for treatment, at a desired anatomical location (cervical carotid artery, for example) in the central circulatory system. The GECKO guidewire itself is not meant to perform a treatment but is used to set the primary access that will allow performance of the treatments.

SUMMARY:
The objective of this clinical investigation is to evaluate the safety and technical success of the Basecamp Vascular controllable directional GECKO guidewire when used to facilitate endovascular access to the targeted vessel in order to treat the vascular lesion.

DETAILED DESCRIPTION:
The Basecamp Vascular trial is a prospective monocenter, non-randomized, open clinical investigation of their controllable directional GECKO guidewire which has not yet received the CE mark. The GECKO active guidewire is a sterile, single-use device to be used by interventional neuroradiologists (INR) to position a distal access catheter (DAC). The device is a system composed of a deflector (the guide) and a handle. The handle contains the battery and integrated electronics. The device can be activated using buttons on the handle. When the user presses a button, a current is transmitted along the guide to its end: this allows the guide to bend (two possible curves). The end of the device can then take an "S" shape. In INR, the placement of a DAC (at the cervical level) is the first step of an endovascular intervention (Primary Access). This is followed by the treatment phase of the vascular pathology with other medical devices (example: embolization, angioplasty). The GECKO active guide is a system that facilitates endovascular navigation and allows the positioning of the DAC via vascular access (femoral or radial artery). The GECKO device is intended to introduce devices used for treatment, at a desired anatomical location (cervical carotid artery, for example) in the central circulatory system. The GECKO guidewire itself is not meant to perform a treatment but is used to set the primary access that will allow performance of the treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years old.
2. An unruptured intracranial aneurysm, a brain arteriovenous malformation (bAVM) or dural arteriovenous fistula (DAVF) or an internal carotid artery (ICA) stenosis.
3. Subject can receive, if necessary, anti-coagulation and anti-platelet therapy according to the standard used in each study center.
4. Subject is eligible to undergo a procedure with the use of contrast media.
5. Subject is willing to comply with protocol requirements and return to the treatment center for all required clinical evaluations and follow-up.
6. Subject has given written informed consent.
7. Life expectancy >12 months.

Exclusion Criteria:

1. Subject is unconscious and unable to directly provide his/her written informed consent.
2. Subject with a type 3 aortic arch will be excluded from the study.
3. Subject is or has been treated with radiation therapy to the neck or chest.
4. Subject has a life-threatening allergy to contrast media (unless treatment for allergy can be tolerated).
5. Subject has a known cardiac disorder, likely to be associated with cardio-embolic symptoms such as atrial fibrillation (AFib).
6. Subject has any condition, which in the opinion of the treating physician, would place the subject at a high risk of embolic stroke.
7. Subject is unable to complete the required follow-up.
8. Subject is pregnant or breastfeeding. (Females of childbearing potential who are less than 45 years old must have a pregnancy test and provide written proof that they are not pregnant prior to inclusion.)
9. Subject has participated in a clinical study within the last 30 days.
10. Subject with cardiac pacemaker or defibrillator.
11. Persons under guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
The cumulative incidence of all adverse events (serious and non-serious) | 30 days
  The cumulative incidence of adverse events (serious and non-serious) related to the non-permanent implanted guidewire device or the procedure occurring from Day 1 to 30 days post-procedure. All Serious Adverse Events will be reported (e.g., any thromboembolic event [intracranial embolus in the targeted vessel territory or other territory, targeted vessel dissection or dissection of any catheterized vessel], major or minor stroke, or death within 30 days of the intervention).

SECONDARY OUTCOMES:
Number of successful GECKO guidewire placements at the target vessels | During procedure
  Technical success is defined as successful navigation, access and correct positioning of the guidewire and the distal access catheter at the target vessel. This will be measured by the number of successful GECKO guidewire placements at the target vessels.
Measurement of the "time" | During procedure
  Measurement of the "time" to navigate the distal access catheter for Primary Access into the target vessel (time from femoral or radial puncture until arrival at the target vessel).
GECKO Procedure Time | During procedure
  Defined as the time measured from the insertion of the GECKO guidewire until the removal of the GECKO guidewire.
Overall Procedure Time | During procedure
  Defined as the time measured from the insertion of the groin or radial access sheath/catheter until the removal of the access sheath
Number of participants with intracranial hemorrhage | 30 Days
  Number of participants with intracranial hemorrhage inclusive of subarachnoid, intraventricular or intraparenchymal hemorrhage (symptomatic).
All-cause mortality. | 30 Days
  All-cause mortality.
Devices Used | During procedure
  All devices used will be recorded as successful or unsuccessful in conjunction with the GECKO guidewire.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Piotin, M.D., Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Background] Brott TG, Halperin JL, Abbara S, Bacharach JM, Barr JD, Bush RL, Cates CU, Creager MA, Fowler SB, Friday G, Hertzberg VS, McIff EB, Moore WS, Panagos PD, Riles TS, Rosenwasser RH, Taylor AJ; American College of Cardiology Foundation; American Stroke Association; American Association of Neurological Surgeons; American College of Radiology; American Society of Neuroradiology; Congress of Neurological Surgeons; Society of Atherosclerosis Imaging and Prevention; Society for Cardiovascular Angiography and Interventions; Society of Interventional Radiology; Society of NeuroInterventional Surgery; Society for Vascular Medicine; Society for Vascular Surgery. 2011 ASA/ACCF/AHA/AANN/AANS/ACR/ASNR/CNS/SAIP/SCAI/SIR/SNIS/SVM/SVS guideline on the management of patients with extracranial carotid and vertebral artery disease: executive summary. A report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines, and the American Stroke Association, American Association of Neuroscience Nurses, American Association of Neurological Surgeons, American College of Radiology, American Society of Neuroradiology, Congress of Neurological Surgeons, Society of Atherosclerosis Imaging and Prevention, Society for Cardiovascular Angiography and Interventions, Society of Interventional Radiology, Society of NeuroInterventional Surgery, Society for Vascular Medicine, and Society for Vascular Surgery. Circulation. 2011 Jul 26;124(4):489-532. doi: 10.1161/CIR.0b013e31820d8d78. Epub 2011 Jan 31. No abstract available. PMID 21282505
- [Background] Lanzino G, Rabinstein AA, Brown RD Jr. Treatment of carotid artery stenosis: medical therapy, surgery, or stenting? Mayo Clin Proc. 2009 Apr;84(4):362-87; quiz 367-8. doi: 10.1016/S0025-6196(11)60546-6. PMID 19339655
- [Result] Jansen O, Szikora I, Causin F, Bruckmann H, Lobotesis K. Standards of practice in interventional neuroradiology. Neuroradiology. 2017 Jun;59(6):541-544. doi: 10.1007/s00234-017-1837-8. Epub 2017 May 19. PMID 28526977
- [Result] Thompson BG, Brown RD Jr, Amin-Hanjani S, Broderick JP, Cockroft KM, Connolly ES Jr, Duckwiler GR, Harris CC, Howard VJ, Johnston SC, Meyers PM, Molyneux A, Ogilvy CS, Ringer AJ, Torner J; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, and Council on Epidemiology and Prevention; American Heart Association; American Stroke Association. Guidelines for the Management of Patients With Unruptured Intracranial Aneurysms: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Aug;46(8):2368-400. doi: 10.1161/STR.0000000000000070. Epub 2015 Jun 18. PMID 26089327
- [Result] Smith TR, Cote DJ, Dasenbrock HH, Hamade YJ, Zammar SG, El Tecle NE, Batjer HH, Bendok BR. Comparison of the Efficacy and Safety of Endovascular Coiling Versus Microsurgical Clipping for Unruptured Middle Cerebral Artery Aneurysms: A Systematic Review and Meta-Analysis. World Neurosurg. 2015 Oct;84(4):942-53. doi: 10.1016/j.wneu.2015.05.073. Epub 2015 Jun 18. PMID 26093360
- [Result] Derdeyn CP, Zipfel GJ, Albuquerque FC, Cooke DL, Feldmann E, Sheehan JP, Torner JC; American Heart Association Stroke Council. Management of Brain Arteriovenous Malformations: A Scientific Statement for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2017 Aug;48(8):e200-e224. doi: 10.1161/STR.0000000000000134. Epub 2017 Jun 22. PMID 28642352
- [Result] Plasencia AR, Santillan A. Embolization and radiosurgery for arteriovenous malformations. Surg Neurol Int. 2012;3(Suppl 2):S90-S104. doi: 10.4103/2152-7806.95420. Epub 2012 Apr 26. PMID 22826821
- [Result] Abbott AL, Paraskevas KI, Kakkos SK, Golledge J, Eckstein HH, Diaz-Sandoval LJ, Cao L, Fu Q, Wijeratne T, Leung TW, Montero-Baker M, Lee BC, Pircher S, Bosch M, Dennekamp M, Ringleb P. Systematic Review of Guidelines for the Management of Asymptomatic and Symptomatic Carotid Stenosis. Stroke. 2015 Nov;46(11):3288-301. doi: 10.1161/STROKEAHA.115.003390. Epub 2015 Oct 8. PMID 26451020
- See also: FDA Executive Summary General Issues: Meeting to Discuss the Evaluation of Safety and Effectiveness of Endovascular Medical Devices Intended to Treat Intracranial Aneurysms — https://www.fda.gov/media/111329/download